CLINICAL TRIAL: NCT05827783
Title: The Effect of Buzzy and Puppet on Pain and Fear During Phlebotomy in Children: A Randomized Controlled Study
Brief Title: The Effect of Buzzy and Puppet on Pain and Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Şeyda BİNAY YAZ, Assistant professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bakircay University
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Pain; Fear; Nurse's Role
Keywords: Pain; Fear; External cold and vibration; pediatrics; Puppet
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study was a randomized controlled experimental study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bee Buzzy (Experimental): Bee Buzzy Group: Bee Buzzy was attached to the 3-6-year-old child included in this group by the researcher on the arm of the nurse to perform the phlebotomy procedure. Bee Buzzy reduces pain thanks to its cold wings and vibration. It helps to distract attention during phlebotomy and reduces the feeling of pain and fear. Bee Buzzy was tied 5 cm above the area from which blood will be drawn, and after waiting for 15 seconds, the nurse performed a phlebotomy.
  Interventions: Procedure: Implementation of Bee Buzzy
- Puppet Zuzu (Experimental): While the nurse was going to perform the phlebotomy operation on the 3-6-year-old child included in this group, one of the researchers (no. 2) tried to distract the child by putting the puppet on her hand and making her talk. The puppet used is an easy-to-use and hand-held puppet that will not cause fear in children. The puppet was named 'Zuzu' by researchers.
  Interventions: Procedure: Implementation of Puppet Zuzu
- Control (No Intervention): No attempt was made to the 3-6-year-old child included in this group, during the process when the nurse performed the phlebotomy. Routine phlebotomy was performed. Pain and fear of the child during the procedure were evaluated.

INTERVENTIONS:
Procedure: Implementation of Bee Buzzy — Implementation of Bee Buzzy It is defined as the use of a device called Bee Buzzy, which applies cold and vibrates in the form of a toy bee, by the researcher for fear and pain during phlebotomy in children.
  Nurse performs phlebotomy on pediatric patients in the pediatric phlebotomy unit. During this application, the researcher puts the Bee Buzzy device on the child's arm just above the area from which blood was taken, and remains attached to the arm during the phlebotomy procedure. This device applies cold and vibrates. Pain and fear during the procedure are evaluated by the researcher, the nurse, and the child's parent.
  Arms: Bee Buzzy
Procedure: Implementation of Puppet Zuzu — Implementation of puppet zuzu It is defined as the use of a puppet that is seized and made to talk by the researcher for fear and pain during phlebotomy in children.
  Nurse performs phlebotomy on pediatric patients in the pediatric phlebotomy unit. During this practice, a puppet is seized by the researcher and made to talk, and the child's attention is tried to be drawn. While this procedure is in progress, the researcher, the nurse, and the child's parent evaluate the pain and fear during the procedure.
  Arms: Puppet Zuzu

SUMMARY:
Summary Aim: This study was conducted to evaluate the effects of the use of Bee Buzzy, external vibrating cold application, and the use of puppets on pain and fear in children aged 3 to 6 years during phlebotomy.

Method: This study is a randomized controlled trial. The study was conducted with 105 children aged 3-6 years who came to the pediatric phlebotomy unit of a university hospital. The sample of children (n=105) was divided into groups (group 1, Bee Buzzy; group 2, puppet; group 3, control) by block randomization. Children's pain and fear scores were evaluated using the Wong-Baker Pain Scale and Child Fear Scale, as well as the investigator's report, after phlebotomy, their parents, and the nurse who attempted phlebotomy.

ELIGIBILITY:
Inclusion Criteria:

* Participants whose child and parents agreed to participate in the study
* Children who had successful phlebotomy on the first attempt

Exclusion Criteria:

* Children with chronic disease, mental disability, or mental retardation
* Children who had taken analgesics in the last 24 hours
* Children who were hospitalized
* Children who had undergone a surgical procedure
* Children who did not have successful phlebotomy on the first attempt

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Statistical difference between groups about pain scores | During the procedure, approximately 5-10 minutes
  Implementation of interventions aimed at reducing pain in experimental groups. Wong-Baker Facial Pain Rating Scale: The Facial Expression Rating Scale is a scale that includes 6 facial expressions and provides a rating between 0-10. This scale, which does not require words, is a reliable and valid measurement tool in the assessment of acute pain. A score of 0 indicates no pain and a score of 10 indicates the highest level of pain. In the scale, it means that as the pain score increases, the pain also increases.
Statistical difference between groups about fear scores | During the procedure, approximately 5-10 minutes
  Implementation of interventions aimed at reducing fear in experimental groups. Children's Fear Scale: This scale includes 5 different facial expressions. This scale is scored between 0-4 and it is stated to be a reliable and valid measurement tool in the evaluation of fear. This scale does not require words. A score of 0 indicates no fear and a score of 4 indicates the highest level of fear. In the scale, it means that as the fear score increases, the fear also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda Binay Yaz, PhD, Principal Investigator — Izmir Bakircay University Hospital
Locations (1):
- Bakırcay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yaz SB, Basdemir S, Gectan E. The effect of vibrating cold application and puppet use on pain and fear during phlebotomy in children: A randomized controlled study. J Pediatr Nurs. 2024 Jan-Feb;74:77-84. doi: 10.1016/j.pedn.2023.11.018. Epub 2023 Nov 28. PMID 38029689